CLINICAL TRIAL: NCT01557218
Title: Increasing the Variety of Vegetables and Fruits Served to Preschool Children at a Snack
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study of Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ChildFood101; R01DK082580 (NIH)
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Obesity; Feeding Behaviors
Keywords: Dietary variety; Vegetable intake; Fruit intake
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Cucumber (Experimental)
  Interventions: Other: Cucumber snack
- Pepper (Experimental)
  Interventions: Other: Pepper snack
- Tomato (Experimental)
  Interventions: Other: Tomato snack
- Vegetable variety (Experimental)
  Interventions: Other: Vegetable variety snack
- Apple (Experimental)
  Interventions: Other: Apple snack
- Peach (Experimental)
  Interventions: Other: Peach snack
- Pineapple (Experimental)
  Interventions: Other: Pineapple snack
- Fruit variety (Experimental)
  Interventions: Other: Fruit variety snack

INTERVENTIONS:
Other: Cucumber snack — Three 300-g bowls of vegetables per table: three of cucumber slices
  Arms: Cucumber
Other: Pepper snack — Three 300-g bowls of vegetables per table: three of yellow pepper strips
  Arms: Pepper
Other: Tomato snack — Three 300-g bowls of vegetables per table: three of grape tomatoes
  Arms: Tomato
Other: Vegetable variety snack — Three 300-g bowls of vegetables per table: one each of cucumber slices, pepper strips, and grape tomatoes
  Arms: Vegetable variety
Other: Apple snack — Three 300-g bowls of fruits per table: three of apple wedges
  Arms: Apple
Other: Peach snack — Three 300-g bowls of fruits per table: three of peach slices
  Arms: Peach
Other: Pineapple snack — Three 300-g bowls of fruits per table: three of pineapple half-rings
  Arms: Pineapple
Other: Fruit variety snack — Three 300-g bowls of fruits per table: of each of apple wedges, peach slices, and pineapple half-rings
  Arms: Fruit variety

SUMMARY:
Intake of vegetables and fruits in preschool children is less than recommended amounts. Although offering a variety of foods has been shown to increase intake, this effect has not been well studied for low-energy-dense foods. The purpose of this study was to test whether increasing the variety of vegetables and fruits served to preschool children affected the amount eaten. The hypotheses were that increasing the variety of vegetables and fruits would increase both the amount selected and the amount eaten.

ELIGIBILITY:
Inclusion Criteria:

* attenders at the relevant child care center

Exclusion Criteria:

* allergy or sensitivity to any test food

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2011-01; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Intake of vegetables and fruit | One month

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. Rolls, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University Laboratory for the Study of Human Ingestive Behavior, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Roe LS, Meengs JS, Birch LL, Rolls BJ. Serving a variety of vegetables and fruit as a snack increased intake in preschool children. Am J Clin Nutr. 2013 Sep;98(3):693-9. doi: 10.3945/ajcn.113.062901. Epub 2013 Jul 31. PMID 23902783